CLINICAL TRIAL: NCT05153421
Title: Clinical Evaluation of the All'InCath CBC 035M When Used for Peripheral Vasculature Percutaneous Transluminal Angioplasty.
Brief Title: Evaluation of All'InCath in Peripheral Vasculature Percutaneous Transluminal Angioplasty.
Acronym: CBC035M
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As part of the new regulatory requirements in Europe and in accordance with the MDR regulation set to take effect on January 1, 2025, NexStep Medical is compelled to prematurely terminate its ongoing clinical study.
Sponsor: NexStep Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-0001
Record Dates: First submitted 2021-10-20; First posted 2021-12-10 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All'InCath CBC 035M Balloon Dilatation Catheter (Experimental): Peripheral Vasculature Percutaneous Transluminal Angioplasty and Control Angiography with single balloon dilatation catheter.
  Interventions: Device: All'InCath CBC 035M Balloon Dilatation Catheter

INTERVENTIONS:
Device: All'InCath CBC 035M Balloon Dilatation Catheter — Peripheral Vasculature Percutaneous Transluminal Angioplasty and Control Angiography with single balloon dilatation catheter.

SUMMARY:
The purpose of this study is to evaluate the clinical safety, performance and benefits (e.g. decrease of procedure time, decrease of radiation time, decrease of the amount of injected contrast, delivery and ease of use) of a novel balloon catheter that combines angiography and angioplasty capabilities.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical safety, performance and benefits (e.g. decrease of procedure time, decrease of radiation time, decrease of the amount of injected contrast, delivery and ease of use) of a novel balloon catheter that combines angiography and angioplasty capabilities when used per its Instructions for Use (IFU) during percutaneous transluminal angioplasty procedures in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide Informed Consent
* Can also be executed by the legal designated representative or the witness
* As per the Principal Investigator's practices as per standard of care, the subject is indicated for PTA in the peripheral vasculature, including iliac, femoral, popliteal, and renal arteries, and any treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistulae.
* Male or female >18 years old.
* Life expectancy >1 year

Exclusion Criteria:

* Unstable coronary artery disease or any other uncontrolled comorbidity.
* Myocardial infarction or stroke within two (2) months before baseline evaluation.
* Previous peripheral bypass or procedure that includes the target vessel.
* Known, untreated allergy or other contraindications to contrast agents or medications used during or after PTA.
* Non-correctable bleeding diathesis, platelet dysfunction, thrombocytopenia, or any other known coagulopathy.
* The use of antiplatelet or anticoagulant therapy is contraindicated.
* Any planned major surgical or interventional procedure within 30 days after the study procedure.
* Females who are breast-feeding or child-bearing potential and not using a medically reliable method of contraception (as defined below) for the entire study duration:
* medically reliable contraception defined as: oral, injectable, or implantable contraceptives, intrauterine contraceptive devices, or those not using another method deemed by the Investigator to be sufficiently reliable.
* subjects who are surgically sterilized / hysterectomized or post-menopausal for longer than two (2) years are not considered childbearing potential.
* Positive pregnancy test result in women of child bearing potential or is breast-feeding.
* Incapacitated individuals and those with psychiatric disorders that could interfere with the provision of informed consent, completion of tests, therapy, follow-up or general study compliance.
* Participation in another study with investigational drug or device within the 30 days preceding and during the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Safety of the All'InCath Contrast Balloon Catheter 035M | immediately post-procedure
  Periprocedural Serious Adverse Events
Performance and effectiveness of the All'InCath Contrast Balloon Catheter 035M | immediately post-procedure
  Vascular patency

SECONDARY OUTCOMES:
Performance of the All'InCath Contrast Balloon Catheter 035M | Time of Procedure
  Duration of the PTA procedure.
Evaluation of the function of the All'InCath Contrast Balloon Catheter 035M | During Procedure
  Investigator opinion
Efficiency and Safety of the All'InCath Contrast Balloon Catheter 035M | During Procedure
  Level of radiation exposure during the PTA (mGy).
Safety and performance of the All'InCath Contrast Balloon Catheter 035M | During Procedure
  Dose of injected contrast medium at the targeted location (mL)
Safety of the All'InCath Contrast Balloon Catheter 035M | 3 days
  Post procedural adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Thaveau, MD, PhD, Principal Investigator — Geprovas
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No